CLINICAL TRIAL: NCT00295269
Title: Late Steroid Rescue Study (LaSRS): The Efficacy of Corticosteroids as Rescue Therapy for the Late Phase of Acute Respiratory Distress Syndrome
Brief Title: Corticosteroids as Rescue Therapy for the Late Phase of Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 355; N01 HR46054; N01 HR46055; N01 HR46056; N01 HR46057; N01 HR46058; N01 HR46059; N01 HR46060; N01 HR46061; N01 HR46062; N01 HR46063; N01 HR46064
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2006-04

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Diseases
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases

INTERVENTIONS:
Drug: Mythylprednisolone

SUMMARY:
The purpose of this study is to assess innovative treatment methods in patients with adult respiratory distress syndrome (ARDS) as well as those at risk of developing ARDS.

DETAILED DESCRIPTION:
BACKGROUND:

ARDS affects approximately 150,000 people in the United States each year. Despite twenty years of research into the mechanisms that cause this syndrome and numerous developments in the technology of mechanical ventilation, the mortality rate has remained greater than 50 percent. In addition to the tragic loss of human life, this condition poses a cost to society because these patients spend an average of two weeks in intensive care units and require multiple high tech procedures. Because of the overwhelming nature of the lung injury once it is established, prevention appears to be the most effective strategy for improving the outlook for those with ARDS.

Basic research has identified numerous inflammatory pathways that are associated with the development of ARDS. Agents that block these mediators prolong survival in animals with lung injury, and a few of them have been tested in human patients. Because of the large number of putative mediators and the variety of ways that their action can be blocked, the possibility for new drug development is almost infinite. This is an exciting prospect, since it envisions the first effective pharmacologic treatment for ARDS. However, preliminary clinical studies have shown conflicting results, and there is an urgent need for a mechanism to efficiently and effectively test new drugs in ARDS. Treatment studies in patients with ARDS are difficult to perform for three reasons. First, the complicated clinical picture makes it difficult to accumulate a large number of comparable patients in any one center. Secondly, there is no agreement on the optimal supportive care of these critically ill patients. Finally, many of the patients meeting study criteria will not be enrolled in study protocols because of the acute nature of the disease process. For these reasons, therapeutic trials in ARDS require multicenter cooperation.

DESIGN NARRATIVE:

This study compared the effect of corticosteroids with placebo in the management of late-phase (greater than seven days) ARDS. The study determined if the administration of the corticosteroid, methylprednisolone sodium succinate, in severe ARDS that was either stable or worsening after seven days, would reduce mortality and morbidity. The primary endpoint was mortality at 60 days. Secondary endpoints included ventilator-free days and organ failure-free days. LaSRS was designed to include 400 patients and began recruiting in the Spring of 1997. In October 1999, the data and safety monitoring board (DSMB) reduced the recruitment target number to 200 patients because the eligible patients were fewer than anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ARDS or has risk factors for ARDS; individuals will be considered at risk if they are critically ill and have trauma, sepsis, shock, pneumonia, inhalation injury, drug overdose, pancreatitis, or hypertransfusion
* Onset of ARDS must be between 7 and 28 days prior to study entry
* Since ARDS onset, bilateral infiltrates must have persisted and participants must have required continuous mechanical ventilation

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1997-03; Study Completion 2005-09

PRIMARY OUTCOMES:
Mortality rates (measured at time of hospital discharge or 60 days after study entry)

SECONDARY OUTCOMES:
Number of ventilator-free days (measured at 28 days following study entry)
Number of organ failure-free days (measured at 28 days following study entry)
Reduction in markers of ongoing inflammation and fibroproliferation (measured at 7 days following study entry)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Abraham, Principal Investigator — University of Colorado, Denver; William Fulkerson, Principal Investigator — Duke University; Leonard Hudson, Principal Investigator — University of Washington; Paul Lanken, Principal Investigator — University of Pennsylvania; Michael Matthay, Principal Investigator — University of California; Alan Morris, Principal Investigator — Latter Day Saints Hospital; David Schoenfeld, Principal Investigator — Massachusetts General Hospital; Henry Silverman, Principal Investigator — University of Maryland; Galen Toews, Principal Investigator — University of Michigan; Arthur Wheeler, Principal Investigator — Vanderbilt University; Herbert Wiedemann, Principal Investigator — The Cleveland Clinic

REFERENCES:
- [Result] Steinberg KP, Hudson LD, Goodman RB, Hough CL, Lanken PN, Hyzy R, Thompson BT, Ancukiewicz M; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network. Efficacy and safety of corticosteroids for persistent acute respiratory distress syndrome. N Engl J Med. 2006 Apr 20;354(16):1671-84. doi: 10.1056/NEJMoa051693. PMID 16625008
- See also: Acute Respiratory Distress Syndrome Clinical Network [ARDSNet] — http://www.ardsnet.org